CLINICAL TRIAL: NCT06619496
Title: Health in Motion- A Digital Fall Prevention Program Designed to be Delivered as a Wraparound Program
Brief Title: Health in Motion Pragmatic Clinical Trial - WRAPAROUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blue Marble Rehab Inc (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Partners In Care Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AG043191-4. v1-wraparound; 2R44AG043191-04A1 (NIH)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: fall; fall prevention; fall injury; fear of falling; fall efficacy

STUDY DESIGN:
Intervention Model Description: comparative prospective observational cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human-led fall prevention programs (Active Comparator): Participants will complete any human-led fall prevention program of their choice, in a group setting either in-person or via Zoom.
  Interventions: Behavioral: Human-led fall prevention program
- Avatar-led fall prevention program (Experimental): Participants will complete an avatar-led fall prevention program at their local community center or community room of their housing complex
  Interventions: Behavioral: Avatar-led fall prevention program

INTERVENTIONS:
Behavioral: Human-led fall prevention program — Human-led evidence-based fall prevention programs include Matter of Balance, Tai Chi Moving for Better Balance, Walk with Ease, or Arthritis Exercise
  Arms: Human-led fall prevention programs
Behavioral: Avatar-led fall prevention program — The avatar-led fall prevention program consists of the Otago Exercise Program
  Arms: Avatar-led fall prevention program

SUMMARY:
Falls among older adults are a serious public health concern, and injuries resulting from falls can cause significant loss of independence, premature death, and higher caregiver burden. Home-based fall prevention programs, such as the Otago Exercise Program, educate older adults about the importance of identifying fall risk and provide strategies for reducing fall risk; however, many are costly and are not scalable, accessible, or sustainable. This project will compare a digital fall prevention program used in a group setting in the community with traditional community-based fall prevention programs.

DETAILED DESCRIPTION:
This study will involve 2 groups. Group 1 will participate in traditional human-led community based fall prevention programs and Group 2 will participate in avatar-led community-based fall prevention program. Metrics of effectiveness include the rate of falls, fall risk, fear of falling, and falls efficacy. Economic benefit will be measured using the European Quality of Life 5-Dimensional Questionnaire, along with hospital and clinical visits. The primary outcome is the incidence of falls (rate in person-months).

ELIGIBILITY:
Inclusion Criteria:

* age of 55 and older
* Score >30 on the TICS (Telephone Interview for Cognitive Screen) or if lower than 30 has assistance to participate

Exclusion Criteria:

* any person who has been told by their physician that they should not exercise

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of falls | change from baseline to end of intervention (about 3 months)
  number of falls during the intervention compared with the self-reported falls at baseline

SECONDARY OUTCOMES:
Timed Up and Go Test | change from baseline to end of intervention (about 3 months)
  Time taken to stand up from a seated position, walk 10 feet, turn around, return to the chair, sit down
4 Stage Balance Test | change from baseline to end of intervention (about 3 months)
  This test measures the ability to stand for 10 seconds in 4 progressively more challenging positions from standing with feet side by side to standing on one leg. The score is equal to the total time taken to achieve the highest level. The maximum score is 40. If a participant is not able to stand with their feet in tandem, they are considered at higher risk of falling.
One Leg Stand Test | change from baseline to end of intervention (about 3 months)
  This test measures the ability to stand for on one leg for up to 30 seconds. If a participant is not able to stand for 5 seconds, they are considered at higher risk of falling.
30 Second Sit to Stand Test | change from baseline to end of intervention (about 3 months)
  This test measures the number of times a participant can stand up from a seated position in 30 seconds.
Fall Risk Questionnaire | change from baseline to end of intervention (about 3 months)
  This is a multi-factorial questionnaire that can be used to predict fall risk. Questions relate to history of falls, gait/balance, muscle weakness, incontinence, sensation/proprioception, depression, vision and medications. The highest (worst) score = 14. A score of 0-3 denotes low fall risk and scores from 4-14 denote higher fall risk.
Activities Specific Balance Confidence Scale (5 level) | change from baseline to end of intervention (about 3 months)
  This questionnaire measures the participant's confidence in performing activities of daily living in which each item is rated from 0% (no confidence) to 100% (complete confidence). It correlates with other measures of self-efficacy and balance measures.
Veteran Rand-12 (VR-12) | change from baseline to end of intervention (about 3 months)
  This questionnaire measures quality of life over the past 4 weeks.
European Quality of Life 5-Dimensional Questionnaire (EQ-5D-5L) | change from baseline to end of intervention (about 3 months)
  This is a standardized measure of health status for clinical and economic appraisal. The test is a self report health state that domains including mobility, self-care, anxiety/depression, pain/discomfort) using a 5 point scale and a visual analog scale (VAS).
Trail Making Test | change from baseline to end of intervention (about 3 months)
  This is a standardized test of cognitive function. The test consists of two Trails, Trail A and Trail B. Trail A requires the participant to tap on 25 numbers on the screen in order from smallest to largest (1, 2, 3, etc). Trail B requires participants to tap on alternative numbers and letters in consecutive order from smallest/first to largest/last (1, A, 2, B, 3, C etc).
modified Fear of Falling Avoidance Behavior Questionnaire (mFFABQ) | change from baseline to end of intervention (about 3 months)
  This is a standardized self-report assessment that measures behaviors that may be avoided due to a fear of falling. The item scores are summed to form a total score ranging from 0 to 56. Higher scores indicate a higher level of fear of falling avoidance behavior
Upstream Social Isolation Risk Scale (USIR-S) | change from baseline to end of intervention (about 3 months)
  A standardized assessment of social isolation. Lower scores indicate lower risk of social isolation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheryl Flynn, Altadena, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared